CLINICAL TRIAL: NCT06551844
Title: Adaptive Dengue Antiviral Platform Trial (ADAPT): a Phase 2 Randomized, Adaptive, Open Label Trial for Antiviral Screening in Patients With Early Symptomatic Dengue
Brief Title: Adaptive Dengue Antiviral Platform Trial
Acronym: ADAPT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 71DX
Record Dates: First submitted 2024-08-06; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Dengue; Antiviral Drugs
MeSH Terms: conditions — Dengue | interventions — molnupiravir

STUDY DESIGN:
Intervention Model Description: This is a phase 2 randomized, adaptive, open label trial for antiviral screening in patients with dengue presenting at the healthcare settings within 48 hours.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (arm A) (No Intervention): Patients, who are randomly allocated into arm A will receive the standard of care (no study drug)
- Molnupiravir (arm B) (Experimental): Patients, who are randomly allocated into arm B, will receive 800mg po bid of Molnupiravir for 5 days
  Interventions: Drug: Molnupiravir 400 mg
- Monoclonal antibody (arm C) (Experimental): Patients, who are randomly allocated into arm C, will receive a single dose of 6mg/Kg of the dengue monoclonal antibody via an intravenous line over 2 hours.
  Interventions: Drug: VIS513 (a monoclonal antibody)

INTERVENTIONS:
Drug: Molnupiravir 400 mg — This is an antiviral drug (an RNA dependent RNA polymerase inhibitor, with broad spectrum antiviral activity) currently approved for use in treatment for COVID-19 patients.
  In this trial, its antiviral effectiveness on the early phase of dengue virus infection will be assessed.
  Other Names: Molnupiravir STELLA 400mg
  Arms: Molnupiravir (arm B)
Drug: VIS513 (a monoclonal antibody) — VIS513 is an engineered humanised monoclonal antibody produced by recombinant DNA technology in a mammalian cell (i.e. Chinese hamster ovary) line. It was discovered in the USA by Visterra Inc and subsequently technology for manufacturing and further development was transferred to Serum Institute of India Pvt. Ltd., Pune, India. It has shown potent, specific neutralization of all four serotypes of DENV.
  Other Names: Dengue monoclonal antibody (Dengue mAb/ Dv Mab)
  Arms: Monoclonal antibody (arm C)

SUMMARY:
This is a randomized, open-label adaptive platform trial aiming to screen the antiviral effectiveness of the experimental drug(s) in early dengue infection

* Primary objectives:

  * To determine the antiviral effectiveness of the experimental drug(s) in early dengue infection
  * To assess the safety and tolerability of the experimental drug(s) in dengue patients
* Secondary objective:

  * To assess the effect of the experimental drug(s) in dengue patients on physiological, clinical and virological parameters

DETAILED DESCRIPTION:
This is a randomized, open-label adaptive platform trial investigating the antiviral effectiveness of various intervention arms in patients with lab-confirmed dengue and less than 48 hours of fever. The antiviral candidates in this trial will include the repurposed antiviral drugs, novel small molecule drugs and dengue monoclonal antibody. Patients will be randomly allocated between available treatment arms and compared to standard of care ("no study drug": no placebos will be made for this trial).

The current sites include Hospital for Tropical Diseases in Ho Chi Minh City, Vietnam. Other sites and countries may be added in due course.

This is a continually running adaptive platform trial, which begins with two initial candidate drugs (a total of 3 arms): molnupiravir and VIS513 (a dengue monoclonal antibody). New therapies may be added and poorly performing arms or interventions meeting pre-specific thresholds for in vivo antiviral efficacy will be removed.

The sample size is adaptive with multiple planned interim analyses. The number of patients recruited depends on the results. For each intervention studied the sample size will be adaptive and determined by pre-specified stopping rules for futility and efficacy. Patients are invited to participate in the trial if they present at the healthcare settings with early symptomatic dengue virus infection (less than 48 hours since the onset of fever and positive NS1 antigen test) and can be able to return for follow up visits at 30 and 60 days after randomization.

The randomization ratios will be uniform for all available and eligible arms (1:1:1...).

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients with a clinical diagnosis of dengue virus infection and less than 48 hours of fever
* Positive NS1 rapid diagnostic test
* >= 10 years or ≥ 18 years of age (depending on license of therapeutic being evaluated)
* Patient is able to give written informed consent or assent for full participation in the study.
* Agreement to stay in hospital for duration of the intervention (most will be 5 days) and follow-up visits at day 30 and 60 post enrolment.

Exclusion Criteria:

* Meets criteria for severe dengue at baseline (severe plasma leakage leading to dengue shock syndrome, fluid accumulation with respiratory distress, severe bleeding, severe organ involvement - AST/ALT>1000 U/L, impaired consciousness, multiple organ dysfunction)
* Pregnancy (either clinically confirmed or by urine dipstick for human chorionic gonadotrophin hormone)
* Breastfeeding women
* Localising features suggesting an alternative/additional diagnosis, e.g. pneumonia, sepsis
* Renal failure (baseline eGFR < 30ml/min)
* History or presence of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, autoimmune, dermatologic or immunosuppressive disorders
* History of allergic disease, allergic reactions or known hypersensitivity to any component of the study product (Mild non-medication allergies allowed)
* Any condition that, in the opinion of the investigator, would complicate or compromise the study or well-being of the participant
* Participation or planned participation in a study involving the administration of an investigational compound within the past one month.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Viral clearance rate | From randomization until day 5 of study
  Rate of viral clearance estimated under a hierarchical log-linear model fit to the serial viral load measurements over 5 days after enrolment. The viremia kinetics will be measured using the qRT-PCR assay, which will be performed on samples taken twice a day from day 1 to day 3 of study and then once a day on days 4 and 5 of study (total 9 samples per patient).
Number of AEs (grade 3, 4 and 5) | Until day 30 post-enrolment
  All patients will be followed up daily until discharge and then at around days 30 after randomization to collect information on clinical progress of dengue illness and any adverse events occurring during the study course. All AEs and SAEs will be recorded.

SECONDARY OUTCOMES:
Area under the viremia curve | From randomisation until day 5 of study
  Area under the curve (AUC) of the serial viremia measurements during the first 5 days of study
Viral log reduction | up to 48 hours of study
  Reduction of viremia at the 24 and 48 hours compared to baseline
NS1 clearance time | up to day 5
  Time to NS1 clearance as estimated under a non-linear model
Number of patients progress to severe dengue (WHO 2009 criteria) | From enrolment until discharge, assessed up to 30 days
  All patients will be followed up daily until discharge to collect information about the clinical progress of dengue
Number of patients requiring for ICU admission | From enrolment until discharge, assessed up to 30 days
  All patients will be followed up daily until discharge to collect information about the clinical progress of dengue
Fever clearance time | From enrolment until discharge, assessed up to 30 days
  Time elapsed from enrolment to the afebrile time-point (defined as body temperature <37.5 °C for at least 48 hours)
Platelet nadir | Until day 30 post-enrolment
  The lowest platelet count recorded during admission
Maximum AST/ALT | Until day 30 post-enrolment
  The highest values of AST/ALT measured
Change in haematocrit | Until day 30 post-enrolment
  Change in haematocrit during the hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Yacoub, MD., PhD., Principal Investigator — University of Oxford, UK
Locations (1):
- Hospital for Tropical Diseases at Ho Chi Minh city, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The database may be shared with researchers not directly involved in this study but only after the main paper has been published and in accordance with OUCRU guidelines on data sharing. The database will only be shared if future publications are not compromised. No identifiable information will be shared with any other person/organisation than that authorised in the protocol.
Supporting Information: Study Protocol
Time Frame: starting 6 months after publications of study findings